CLINICAL TRIAL: NCT06018831
Title: Urine and Ultrasound Screening for Kidney Disease in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Kunshan City Maternal and Child Health Hospital (Unknown); Qidong City Maternal and Child Health Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2021YFC2500202
Record Dates: First submitted 2023-02-03; First posted 2023-08-31 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Kidney Diseases; Diagnostic Techniques; Ultrasound; Urinalysis; Child, Only
MeSH Terms: conditions — Kidney Diseases | interventions — Urination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urine and Ultrasound Screening (Experimental): About 10,000 children called KunQi Cohort are born in Jiangsu Province(8,000 in Kunshan and 2,000 in Qidong) and about 3,000 born in Shanghai. Children will receive urine and ultrasound screening in 0-3 months ,and complete 3 to 6 years of follow-up( at least one type screening every year)
  Interventions: Other: Urine and Ultrasound Screening

INTERVENTIONS:
Other: Urine and Ultrasound Screening — When an infant was born, he/she will receive the first urine and ultrasound screening in 3 months in Kunshan/Qidong City Maternal and Child Health Hospital.In Kunqi Cohort, 9,000 will complete 3 years follow-up(urine screening once every year, another ultrasound screening in 24-30 months). Urine sample (50ml) will be stored only once within one year. Dry blood filter paper(120ul) will be stored once a year when he or she has a blood routine for future study.1,000 children will complete 6 year follow-up(receive urine and ultrasound screening once every year). Urine sample (50ml) will be stored once a year. Dry blood filter paper(120ul) will be stored once a year when he or she has a blood routine for future study. The 14 urine test items include: leukocytes, urobilinogen, microalbumin, protein, bilirubin, glucose, ascorbic acid, specific gravity, ketone bodies, nitrite, creatinine, pH, occult blood, and urinary calcium. Ultrasound test will screen for kidneys, ureters and the bladder.

SUMMARY:
The aim of this study is to early detect kidney disease in the natural population cohort of children by urine and ultrasound screening, to assist in the precise prevention and treatment of children's kidney disease, and to establish a risk prediction system for children's kidney disease. About 10,000 children called KunQi Cohort are born in Jiangsu Province(8,000 in Kunshan and 2,000 in Qidong) and about 3,000 born in Shanghai. Through the project, child who is found with abnormal urine or ultrasound result will be referred to Children's Hospital of Fudan University to get further examination and treatment.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) often has an insidious onset. Early detection of CKD and more aggressive treatment and monitoring of high-risk CKD patients at risk of progression are the consensus of current medical practice. However, there is currently no CKD risk prediction system for the Chinese population, especially children. The main goal of this project is to establish a risk prediction system for children's kidney disease, and to assist in the precise prevention and treatment of children's kidney disease. The project is based on the "urine and ultrasound screening" strategy that has been carried out for more than ten years in Shanghai, using a non-invasive and effective screening method in the natural population cohort of children, in order to detect kidney disease in the early stage.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive live newborn infants(regardless of physical condition)
* Complete at least 3 years of follow-up

Exclusion Criteria:

* Declining the screening
* Missing

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13000 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence, incidence, and incidence of renal disease progression in children with CKD | From baseline to the third or sixth year of the study
  The number of CKD patients diagnosed according to the routine diagnosis and treatment of the department of nephrology in Children's Hospital of Fudan University in the 3-6 year observation period accounted for the percentage of the total cases studied.

SECONDARY OUTCOMES:
Urine metabolomic and proteomic profiles in KunQi Cohort | From baseline to the third or sixth year of the study
  9,000 children's urine samples (50ml) will be stored as biospecimen retention at -80°C only once within one year, another 1,000 children's urine samples (50ml) will be stored also as biospecimen retention at -80°C once a year.
  Biospecimen retention will be used to characterize the urinary and metabolome and proteome in children also expect to identify urine biomarkers for the early diagnosis of CKD.
Blood metabolomic and DNA profiles in KunQi Cohort | From baseline to the third or sixth year of the study
  Dry blood filter paper(120ul) will be stored once a year when he or she has a blood routine for metabolomic study and DNA extraction, aiming to identify blood metabolomic biomarkers and DNA mutations for the early diagnosis of CKD.
Potential risk factors asked within questionnaire for the onset, development and prognosis of CKD in children | From baseline to the third or sixth year of the study
  Every child's patient will be asked to complete 3-6 year follow-up questionnaire once a year(include Children Kidney Health Survey for first-year baseline questionnaire and Chilren Kidney Health Survey as every year's follow-up questionnaire) when undergoing routine child health checkups, which includes health conditions and kidney disease related events including family history, mother's height and weight before and after pregnancy (used to calculate BMI), parents' smoking and drinking history, whether the mother takes antihypertensive drugs and the type, parents' occupational exposure history, drinking water quality, take-out frequency, mother's first child bearing age and the age of this child bearing, newborn hospitalization history. These potential risk factors analyzed by statistical methods are aimed to predict the onset, development and prognosis of CKD in children.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Qidong City Maternal and Child Health Hospital, Nantong, Jiangsu
  - Kunshan City Maternal and Child Health Hospita, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gong Y, Zhang Y, Shen Q, Xiao L, Zhai Y, Bi Y, Shen J, Chen H, Li Y, Xu H. Early detection of congenital anomalies of the kidney and urinary tract: cross-sectional results of a community-based screening and referral study in China. BMJ Open. 2018 May 30;8(5):e020634. doi: 10.1136/bmjopen-2017-020634. PMID 29848771
- [Background] Gong Y, Xu H, Li Y, Zhou Y, Zhang M, Shen Q, Huang J, Xu H, Bi Y, Chen H, Zhang Y, Wang J. Exploration of postnatal integrated management for prenatal renal and urinary tract anomalies in China. J Matern Fetal Neonatal Med. 2021 Feb;34(3):360-365. doi: 10.1080/14767058.2019.1608176. Epub 2019 Apr 29. PMID 30983458
- [Background] Zhai YH, Xu H, Zhu GH, Wei MJ, Hua BC, Shen Q, Rao J, Ge J. Efficacy of urine screening at school: experience in Shanghai, China. Pediatr Nephrol. 2007 Dec;22(12):2073-9. doi: 10.1007/s00467-007-0629-5. Epub 2007 Oct 18. PMID 17943322
- [Derived] Shen Y, Liu T, Liu J, Han X, Wu J, Xie L, Chen X, Xu B, Sun Y, Xu S, Zhang Q, Xie N, Zhang L, Ji J, Mo W, Liu Y, Shi X, Shen J, Qiu W, Huang J, Shen Q, Zhai Y, Xu H; KQBC group. Kun-Qi birth cohort (KQBC) study for the incidence, aetiology and risk factors of chronic kidney disease in Chinese children: a cohort profile. BMJ Open. 2025 Aug 16;15(8):e102702. doi: 10.1136/bmjopen-2025-102702. PMID 40819875